CLINICAL TRIAL: NCT03827486
Title: EFFECTIVENESS OF A PROGRAM OF DOMICILIARY EXERCISES AGAINST HABITUAL CLINICAL PRACTICE IN THE RECURRENCE OF ACUTE LOW BACK PAIN: RANDOMIZED CLINICAL TRIAL
Acronym: LUMBAREX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Rossana Chiesa Estomba, MD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUMBAREX
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Standard of Care; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator)
  Interventions: Other: Standard of care (exercise)
- Domicilary exercise program (Experimental)
  Interventions: Other: Domicilary exercise program

INTERVENTIONS:
Other: Standard of care (exercise) — Exercise program according to the standard of care
  Arms: Standard of care
Other: Domicilary exercise program — Domicilary exercise program according to protocol (evidence based medicine)
  Arms: Domicilary exercise program

SUMMARY:
Introduction: Low back pain is a frequent and universally distributed symptom that affects people of any age and both sexes. Approximately 80% of the population will present it at some point in their life. Acute low back pain lasts less than 4 weeks, subacute 4 to 12 weeks and chronic more than 12 weeks.

Hypothesis: Treatment with an exercise program combined with the usual treatment decreases the recurrence of acute low back pain, as well as improvements in pain, functionality, and quality of life of patients.

Principal Objective To evaluate the decrease of recurrence of low back pain in the medium-long term of the patients who perform an exercise program compared to those who do not, with both groups receiving the same pharmacological treatment and information of the postural hygiene guidelines endorsed by the current scientific societies.

Methods: Patients between 18 and 65 years of age who come to the emergency room with acute low back pain and who meet the eligibility criteria proposed for this study. At the first visit, patients in a control group and intervention group will be randomized. Pharmacological treatment and postural hygiene guidelines will be indicated for both groups, adding the exercise table to the intervention group. The variables chosen are the questionnaires Oswestry for functionality, Goldberg, EuroQol-5D for the quality of life, and VAS for pain; which will be measured in the first consultation, at one month, at three and at six months.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old.
2. Low back pain of non-traumatic origin.
3. Signature of informed consent.
4. Availability for compliance with the intervention and commitment to send the study questionnaires.
5. A correct domain of the Spanish language.

Exclusion Criteria:

1. Pregnant women and breastfeeding
2. Any underlying pathology that contraindicates the use of the drugs (NSAIDs, paracetamol) included in this study.
3. Rheumatological diseases that cause spinal involvement (e.g., spondyloarthritis)
4. Low back pain with clinical or associated neurological deficit
5. History of active cancer or remission less than one year
6. Pathological previous image test that shows a causal relationship with the episode under study (e.g. fracture-vertebral crush, herniated disc, etc.)
7. Low back pain associated with other systemic pathologies (eg urinary infection, retroperitoneal hematomas, pancreatitis, etc.)
8. Fever
9. Patients with usual analgesic treatment superior to the 1st step of WHO.
10. Major psychiatric pathology diagnosed not stable (pharmacological treatment not stable in the last 6 months) except depression
11. Neuromuscular pathology diagnosed
12. Having some of the following diseases: fibromyalgia, chronic fatigue syndrome, chronic low back pain diagnosed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who present a new process | 3 months
  Patient who present a recurrence

IPD SHARING:
Plan to Share IPD: No